CLINICAL TRIAL: NCT02030756
Title: Assessment of the Performance, Efficacy and Safety of Vibrating Capsule Medical Device in Aiding Reliving Constipated Individuals.
Brief Title: Performance, Efficacy and Safety of Vibrating Capsule in Aiding Constipated Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vibrant Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Vibrant-14-MS-CTIL
Record Dates: First submitted 2014-01-07; First posted 2014-01-08 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Chronic Idiopathic Constipation
Keywords: constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vibrating capsule (Active Comparator): patients will receive vibrating capsule for 8 weeks of treatment [1 every 3 days (+/- 1 day)].
  Interventions: Device: vibrating capsule
- sham non-vibrating capsule (Sham Comparator): patients will receive sham non-vibrating capsule for 8 weeks of treatment [1 every 3 days (+/- 1 day)].
  Interventions: Device: sham non-vibrating capsule

INTERVENTIONS:
Device: vibrating capsule — patients will receive vibrating capsule for 8 weeks of treatment [1 every 3 days (+/- 1 day)].
  Arms: Vibrating capsule
Device: sham non-vibrating capsule — patients will receive sham non-vibrating capsule for 8 weeks of treatment [1 every 3 days (+/- 1 day)].
  Arms: sham non-vibrating capsule

SUMMARY:
This is a study intended to evaluate the efficacy and safety of the vibrating capsule versus sham non-vibrating capsule on spontaneous bowel movement, in aiding reliving Constipated Individuals

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years and older.
2. Patients with chronic idiopathic constipation according to Rome III criteria and who have not experienced relief of their symptoms from available therapies (osmotic and stimulant laxatives which was used for at least one month at recommended dose).
3. Patients with more than 1 bowel movement/2 weeks and < 3 bowel movement/week.
4. Colonoscopy performed in the past 10 years prior to study participation, unless the patients are <50 years old and without alarming signs and symptoms
5. Patient signed ICF
6. For women with childbearing potential, adequate contraception

Exclusion Criteria:

1. History of complicated/obstructive diverticular disease
2. History of intestinal or colonic obstruction.
3. History of significant GI disorder.
4. Use of following medication: Medication that may affect the bowel mobility, Prokinetics, Anti-Depressants, medications for treatment of Parkinson disease, Opiates, Calcium-channel Blockers, Aluminium/Magnesium Hydroxids
5. Clinical evidence of significant respiratory, CVS, renal, hepatic, biliary, endocrine, psychiatric, neurologic, or presence of abdominal pacemakers.
6. Presence of pacemaker.
7. History of, or current eating disorders, such as anorexia, bulimia, or compulsory overeating.
8. Diagnosis of mega-rectum or colon, a history of intestinal obstruction, congenital anorectal malformation, clinically significant rectocele, or any evidence of intestinal structural abnormality, including GI resection that affects bowel transit, or any evidence of intestinal carcinoma or inflammatory bowel disease of alarm symptoms such as weight loss, rectal bleeding, or anaemia.
9. History of Zenker's diverticulum, dysphagia or a known esophageal stricture 10. Chronic use of non-steroidal anti-inflammatory drugs (NSAIDs)

11. Participation in another clinical study in the last 4 months prior to screening.

12. Any other condition which in the opinion of the investigator may adversely affect the safety of the patient or would limit the patient's ability to complete the clinical study.

13. Women who are pregnant or lactating.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Frequency of bowel movements | 3 months
  change from baseline in the weekly Spontaneous Bowel Movement (SBM) rate during treatment period. Success will be defined as increase by at least 1 SBM/week. The primary analysis will be a comparative analysis of success rates between the study groups

CONTACTS AND LOCATIONS:
Locations (18):
- United States (11):
  - Borland-Groover Clinic, Jacksonville, Florida
  - Georgia Regents University, Augusta, Georgia
  - MGG Group Co., Inc., Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Mgh Boston, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Albuquerque Neuroscience, Albuquerque, New Mexico
  - NYU Langone Medical Center, New York, New York
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - CTRS LLC, Pittsburgh, Pennsylvania
  - Huoston Methodist Hosptial, Houston, Texas
- Israel (7):
  - Bat-Yamon, Bat Yam
  - Degani center Clalit MC, Hadera
  - Expert clinic Clalit MC, Herzliya
  - Talpiot clinic Clalit MC, Jerusalem
  - Zvoulon MC Clalit MC, Kiryat Bialik
  - 100 Tower, Tel Aviv
  - Souraski Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: Yes